CLINICAL TRIAL: NCT03525951
Title: Parent-Level Predictors of Early Language Interaction Quality and Intervention Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-0405; 1K23DC017763-01A1 (NIH); L&S/COMMUN SCI & DISORDERS (Other: UW Madison); Protocol version 2/25/25 (Other: UW Madison)
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Language Development Disorders; Autism Spectrum Disorder
MeSH Terms: conditions — Language Development Disorders; Autism Spectrum Disorder

STUDY DESIGN:
Intervention Model Description: Study 1 (Remote) : Participants in the TD and DLD groups will receive no treatment; observational data only.
  Study 2 (Remote): Participants in the DLD and ASD+DLD groups will receive the Enhanced Milieu Teaching intervention. Participants in the TD will serve as the no-treatment comparison group.
Who Masked: Outcomes Assessor
Masking Description: The research team members doing the language sample analysis and behavioral coding will be blind to group membership (Study 1 and 2) and whether the session was recorded pre-test vs. posttest (Study 2).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Typically Developing Children Study 2 (TD2) (Other): No-intervention comparison group measured over time.
  Interventions: Other: no intervention comparison group
- Children with Dev Language Disorder Study 2 (DLD2) (Experimental): Enhanced Milieu Teaching
  Interventions: Behavioral: Enhanced Milieu Teaching
- Children with Autism Spectrum Disorders Study 2 (ASD+DLD 2) (Experimental): Enhanced Milieu Teaching
  Interventions: Behavioral: Enhanced Milieu Teaching
- Typically Developing Children Study 1 (TD1) (Other): No-intervention group for observational data comparison.
  Interventions: Other: no intervention comparison group
- Children with Dev Language Disorder Study 1 (DLD1) (Other): No-intervention group for observational data comparison.
  Interventions: Other: no intervention comparison group

INTERVENTIONS:
Behavioral: Enhanced Milieu Teaching — The parent training will incorporate the EMT strategies of responsive interaction, matched turns, language modeling, and expansions. There will be three, hour-long parent training sessions following the teach-model-coach-review format (TMCR). The TMCR framework teaching component will involve 10 minutes of verbal and visual instruction on the language stimulation target of interest. The teaching component will be followed by 15 minutes of clinician modeling of the target strategies with the child while the parent watches. The parent will then have the opportunity to practice using the strategy during naturalistic interaction with their child. The clinician will provide individualized coaching on the use of the target strategy during this 20-minute, parent-child interaction. Finally, the clinician will review the target strategies and set goals.
  Arms: Children with Autism Spectrum Disorders Study 2 (ASD+DLD 2); Children with Dev Language Disorder Study 2 (DLD2)
Other: no intervention comparison group — No intervention for observational (Study 1 and 2) and training (Study 2) data comparison.
  Arms: Children with Dev Language Disorder Study 1 (DLD1); Typically Developing Children Study 1 (TD1); Typically Developing Children Study 2 (TD2)

SUMMARY:
Children with poor early language skills are at risk for academic, social, vocational, and health difficulties across the lifespan. Parent training-as part of early language intervention-is a cost-effective option to address this public health issue, but these interventions demonstrate large individual differences in outcomes and barriers to scalability. The purpose of this research is to examine parent-level predictors of early language interaction quality and modifiability during training, which will help increase intervention effectiveness.

DETAILED DESCRIPTION:
This is a minimal-risk, behavioral clinical trial for adult parents and their children (2;6-4;0). The purpose of this study is to determine if and how parent language skills and behavioral awareness influence early language interactions and parent training. Participants will include parent-child dyads in three groups: 1) children who are typically developing (TD; Study 1 and 2), 2) children at risk for persistent developmental language disorder (DLD; Study 1 and 2), and 3) children with autism spectrum disorder and at risk for persistent DLD (ASD+DLD; Study 2). The investigators will examine whether parental language skills predict early language interaction quality (Aim 1; Study 1), whether parental behavioral awareness predicts modifiability during training (Aim 2; Study 2), and whether these predictors vary across children-specifically TD children, children with DLD, or with ASD+DLD (Aim 3; Study 2). The primary outcome measure will be parents' use of language stimulation strategies. The secondary outcome measure will be the number of adult-child conversational turns. The investigators hypothesize that parent language skills (Study 1) and behavioral awareness (Study 2) will be positively associated with the outcomes. However, the strength of the association may vary across the groups. The Study 1 protocol will involve a screening session and observational data collection sessions (TD and DLD groups). Study 1 will be a fully remote model of data collection. The Study 2 protocol will involve five sessions-baseline data collection (all groups), three parent training sessions (DLD and ASD+DLD), and follow-up data collection (all groups) across approximately five weeks. Study 2 will be fully remote. The investigators will collect data from demographic questionnaires, language and learning assessments, measures of parental behavioral awareness, and measures of parent-child language interaction quality (Study 1 and 2). These measures will be administered before and after three parent training sessions (Study 2). These sessions will follow the Teach-Model-Coach-Review framework (TMCR; 1) to train the Enhanced Milieu Teaching (EMT) strategies of responsive interaction, matched turns, language modeling, and expansions. After the training, parent-child dyads will complete the structured interaction and behavioral awareness tasks again (Study 2). The investigators will conduct inter- and intra-group analyses to explore the relationships between the independent (i.e., parent language abilities and behavioral awareness) and dependent (i.e., parent-child language interaction quality and parent modifiability during training) variables.

ELIGIBILITY:
Inclusion - Parents

* Live in a Pennsylvania or New Jersey zip code that is within a 30-mile radius of Weiss Hall at Temple University (STUDY 1) or live in Wisconsin (STUDY 2).
* Have access to the internet and willingness to videoconference (STUDY 1 AND 2)

  a. If a family does not have an adequate digital device (e.g., smartphone only) to videoconference and complete testing, we might lend them a device.
* 18 or older (STUDY 1 AND 2)
* Be an adult parent able to consent for the child to participate in the study (parents in this study can include any caregiver who meets these criteria) (STUDY 1 AND 2)
* English dominant (at least 80%) (STUDY 1 AND 2)
* Have no self-reported diagnosed hearing loss (or no concerns if they have not been tested) (STUDY 1 AND 2).
* Have no reported disabling developmental or acquired disorders or impairments that might significantly affect their performance beyond autism spectrum disorder (ASD) or speech-language disorders (e.g., legal blindness, Down Syndrome, traumatic head injury, stroke) (STUDY 1 AND 2).

Inclusion - Children, Typically Developing Group (TD) (Study 1 and 2)

* age 1 year 4 months - 1 year 8 months 30 days at the start of testing
* English dominant (at least 80%)
* No parent-reported diagnosed hearing loss (or no concerns if the child has not been tested).
* Have typical language abilities as evidenced by meeting two criteria:

  1. Score above the 10th percentile on the Mac Arthur Communicative Development Inventories-Words and Sentences (CDI-WS; long form) Complexity section using sex-specific norms.
  2. Score above the 10th percentile on the CDI-WS (long form) Words Produced using sex-specific norms
* Meet cognitive inclusion criteria: Score greater than or equal to 81.25 standard score (-1.25 SD) on the Cognition subtest of the DAYC-2
* Have no parent reported disabling developmental or acquired disorders/impairments that might significantly affect their performance including speech- language disorders (e.g., ASD, DLD, cancer, stroke, legal blindness, intellectual disability, Down Syndrome, traumatic head injury, cerebral palsy, seizures, or a genetic condition associated with neurodevelopmental disability).
* Pass the Modified Checklist for Autism in Toddlers-Revised with Follow-Up screener

Inclusion - Children, DLD Group (study 1 and 2)

* age 2 years 6 months - 4 years 0 months 0 days at the start of testing
* English dominant (at least 80%)
* No parent-reported diagnosed hearing loss (or no concerns if the child has not been tested).
* Qualify as at risk for persistent language disorder by meeting two criteria:

  1. Score at or below the 10th percentile on the Mac Arthur-Bates Communicative Development Inventory-III (CDI-III) Sentences section using sex-specific norms. For children over 37 mos., score must be less than or equal to the 10th percentile equivalent for 37 mos.
  2. Score at or below the 10th percentile on the CDI-III Vocabulary section using sex-specific norms. For children over 37 mos., score must be less than or equal to the 10th percentile equivalent for 37 mos. The child must also produce at least 10 different words on either the CDI-III or CDI-Words and Sentences (CDI-WS long form).
* Meet cognitive inclusion criteria: Score greater than or equal to 70 standard score (-2 SD) on the Cognition subtest of the DAYC-2 (Voress et al., 2012).
* Have no parent reported disabling developmental or acquired disorders/impairments that might significantly affect their performance beyond speech- language disorders (e.g., ASD, cancer, stroke, legal blindness, intellectual disability, Down Syndrome, traumatic head injury, cerebral palsy, seizures, or a genetic condition associated with neurodevelopmental disability other than DLD).
* Pass the Modified Checklist for Autism in Toddlers-Revised with Follow-Up screener

Inclusion - Children, DLD+ASD Group (STUDY 2)

* 2 years 6 months - 4 years 0 months 0 days at the start of testing
* English dominant (at least 80%)
* No parent-reported diagnosed hearing loss (or no concerns if the child has not been tested).
* Have received ASD diagnosis from a healthcare professional prior to beginning the study.
* Qualify as at risk for persistent language disorder by meeting two criteria:

  1. Score at or below the 10th percentile on the Mac Arthur-Bates Communicative Development Inventory-III (CDI-III) Sentences section using sex-specific norms.

     For children over 37 mos., score must be less than or equal to the 10th percentile equivalent for 37 mos.
  2. Score at or below the 10th percentile on the CDI-III Vocabulary section using sex-specific norms. For children over 37 mos., score must be less than or equal to the 10th percentile equivalent for 37 mos. The child must also produce at least 10 different words on either the CDI-III or CDI-Words and Sentences (CDI-WS long form).
* Meet cognitive inclusion criteria: Score greater than or equal to 70 standard score (-2 SD) on the Cognition subtest of the DAYC-2 (Voress et al., 2012).
* Have no parent reported disabling developmental or acquired disorders/impairments that might significantly affect their performance beyond speech-language disorders or ASD (e.g., cancer, stroke, legal blindness, intellectual disability, Down Syndrome, traumatic head injury, cerebral palsy, seizures, or a genetic condition associated with neurodevelopmental disability other than ASD/DLD).

Min Age: 30 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2025-09-18 (Actual); Study Completion 2025-09-18 (Actual)

PRIMARY OUTCOMES:
Parental Language Stimulation Strategies (Study 2; Remote) | Baseline to Post-treatment (Five Weeks)
  The investigators will code the structured interaction task for parents' use of language stimulation strategies.The investigators will code use of trained strategies (i.e., responsive interaction, matched turns, language modeling, and expansions) and untrained generalization measures like constructive directives and scaffolds. This primary outcome will be a composite score of these language stimulation strategies (e.g., responsive interaction, matched turns, language modeling, expansions, constructive directives, and scaffolds). This composite will be measured at baseline and post-treatment during the structured interaction task, so the same amount of time will be given to each participant to interact. This is a continuous outcome variable, with values greater than or equal to zero. Higher values are generally representative of higher-quality language interactions.
Parental Language Stimulation Strategies (Study 1; Remote) | Baseline (Single Timepoint)
  The investigators will code the structured interaction task for parents' use of language stimulation strategies.The investigators will code use of trained strategies (i.e., responsive interaction, matched turns, language modeling, and expansions) and untrained generalization measures like constructive directives and scaffolds. This primary outcome will be a composite score of these language stimulation strategies (e.g., responsive interaction, matched turns, language modeling, expansions, constructive directives, and scaffolds). This composite will be measured once during the structured interaction task, so the same amount of time will be given to each participant to interact. This is a continuous outcome variable, with values greater than or equal to zero. Higher values are generally representative of higher-quality language interactions.

SECONDARY OUTCOMES:
Adult-Child Conversational Turns (Study 2; Remote) | Baseline to Post-treatment (Five Weeks)
  The investigators will code the number of adult-child conversational turns during the structured language interactions. These turns will be measured at baseline and post-treatment during the structured interaction task, so the same amount of time will be given to each participant to interact. This is a continuous outcome variable, with values greater than or equal to zero. Higher values are generally representative or higher-quality language interactions.
Adult-Child Conversational Turns (Study 1; Remote) | Baseline (Single Timepoint)
  The investigators will code the number of adult-child conversational turns during the structured language interactions. These turns will be measured once during the structured interaction task, so the same amount of time will be given to each participant to interact. This is a continuous outcome variable, with values greater than or equal to zero. Higher values are generally representative or higher-quality language interactions.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca M Alper, Ph.D., CCC-SLP, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make every effort to share the data and findings widely within the allowances of human subjects and other relevant regulations. The study protocol and deidentified data will be made available via clinicaltrials.gov in accordance with those policies. Dr. Alper is an approved PI through Databrary-a secure video data library for behavioral scientists. Participants will have the opportunity to consent to share their data with other approved researchers on Databrary. A variety of permission levels are allowed through Databrary (e.g., solely for approved researchers, for educational and research purposes, etc.).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: All tasks (e.g., the behavioral awareness assessment), protocols (e.g., the parent-child interaction coding), and other research products developed as part of this study will be made available to other researchers upon request after publication of the findings.The parent-child interaction videos and deidentified data that have been released for Databrary will be shared to the repository after the publication of the findings. The consent form will be uploaded within 60 days of the last study visit. The analysis plan will be uploaded with the final results.
Access Criteria: Described above.

DOCUMENTS (1):
  • Informed Consent Form (2024-03-05): https://cdn.clinicaltrials.gov/large-docs/51/NCT03525951/ICF_000.pdf